CLINICAL TRIAL: NCT06514196
Title: Post- Approval Study 1: Long Term Follow Up of the Hintermann Series H® Total Ankle Replacement System
Brief Title: Post- Approval Hintermann Series H® Study 1
Status: Active, not recruiting | Type: Observational
Sponsor: DT MedTech, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PAS 001
Record Dates: First submitted 2024-06-20; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Ankle Osteoarthritis; Post-Traumatic Osteoarthritis of Ankle; Osteoarthritis of Ankle Secondary to Inflammatory Arthritis (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Hintermann Series H3 Total Ankle Replacement System — The H3 includes a metal tibial component, a polyethylene sliding insert (PE inlay), and a metal talar component.

SUMMARY:
The H3 TAR device received U.S. Food and Drug Administration (FDA) Premarket Approval (PMA) on June 4, 2019, and as a condition of that approval, this study is being conducted to provide long-term safety and effectiveness of the H3 TAR System among patients included in the Primary Safety and Effectiveness (PSE) Cohort (P1600361).

This will be a Prospective, single-center, single arm study.

DETAILED DESCRIPTION:
The Hintermann Series H3® (H3) prosthesis is a mobile bearing total ankle replacement (TAR) indicated for use as a non-cemented implant to replace a painful arthritic ankle joint due to primary osteoarthritis, post-traumatic osteoarthritis or arthritis secondary to inflammatory disease (e.g., rheumatoid arthritis, hemochromatosis, etc.).

This will be a Prospective, single-center, single arm study. All living subjects who participated in the PSE cohort, regardless of whether or not the subject has had a revision/removal followed through the 10-year post-operation visit. 298 subjects were originally included in the PSE cohort.

Through 10 years follow up. Based on the last surgery date, it is projected the study will be completed with the final 10-year follow-up visit to occur in December 2024.

Patients will undergo clinical and radiographic evaluation at 5 and 10 years (+/- 90 days) post-operation.

Performance Goals (PGs) will be constructed for the 10-year endpoint. As with the PGs used in the PMA study, these will be based on a prospectively defined, systematic meta-analysis of available published literature and registry data for the control (a legally marketed mobile bearing ankle). The details of the meta-analysis will be pre-specified in a protocol for this purpose. Both the protocol and the meta-analysis will be completed prior to the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Primary diagnosis of osteoarthritis, post-traumatic arthritis or rheumatoid arthritis
* Primary total ankle replacement
* Unilateral or the first ankle implanted if bilateral and the surgery dates for both sides are at least 6 months apart
* Implanted with the correct device without screws (for investigational arm),
* 3rd generation Hintermann Series H3 Total Ankle Replacement;
* Poor pre-operative American Orthopaedic Foot and Ankle Society Hindfoot Score (< 60 points)
* Implanted in 2013 or earlier). Note that all subjects implanted in 2013 or earlier were included regardless of whether they were revised prior to the 2 year endpoint.
* Gave informed consent (unless IRB/Ethics Committee waived this requirement)

Exclusion Criteria:

* Prior TAR or arthrodesis at the involved ankle joint

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all living subjects who participated in the PSE cohort, regardless of whether or not the subject has had a removal/revision followed through the 10-year post-operation visit.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
AOFAS Score Measurement | 10 Years
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score is among will be used for measuring the outcome of treatment in patients who sustained a complex ankle or hindfoot injury. It will be measured at a minimum 10 years post-operation
Survivorship Measurement | 10 Years
  Survivorship (absence of removal/revisions to include polyethylene revision) will be recorded at 10 years from surgery
Serious device-related adverse event Measurement | 10 Years
  Percentage of subjects with a serious device-related adverse event, other than a revision or removal will be calculated at 10 years from surgery
Reoperation, revisions or removals Measurement | 10 Years
  Safety Reporting of the reoperation, revisions or removals of the Hintermann Ankle device will be reviewed and analyzed
Serious Device-Related Adverse Events Measurement | 10 Years
  Incidence, occurrence, and types of serious device-related adverse events will be reviewed and analyzed for subjects Nature, onset, duration, severity, relationship to the device, and relationship to the operative procedure and outcome of any adverse event will be measured.
Device Explant Analysis Measurement | Through Study Completion an Average of 10 years
  Any explanted devices / device components will be returned and handled for analysis as described in Attachment G: Explant and Revision Protocol, to be examined for wear and damage.

CONTACTS AND LOCATIONS:
Overall Officials: Beat Hintermann, Principal Investigator — Cantonal Hosptal, Baselland
Locations (1):
- Kantonsspital Baselland, Bruderholz, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided